CLINICAL TRIAL: NCT02728453
Title: SGLT2 Inhibition With Empagliflozin in Patients With Type 2 Diabetes Mellitus: Influences on Left Ventricular Mass, Function, and Cardiac Lipid Content
Brief Title: SGLT2 Inhibition and Left Ventricular Mass
Acronym: EMPATROPHY
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient recruitment.
Sponsor: Hannover Medical School (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRC-KliPha-001
Record Dates: First submitted 2016-03-24; First posted 2016-04-05 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Empagliflozin (Experimental): 25 mg/d empagliflozin + matching glimepiride placebo for 24 weeks.
  Interventions: Drug: Empagliflozin
- Glimepiride (Active Comparator): 2 or 4 mg/d glimepiride+ matching empagliflozin placebo for 24 weeks.
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Empagliflozin — Treatment with empagliflozin vs. glimepiride to understand whether empagliflozin may reduce left ventricular mass in patients with type 2 Diabetes mellitus.
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Glimepiride — Treatment with empagliflozin vs. glimepiride to understand whether empagliflozin may reduce left ventricular mass in patients with type 2 Diabetes mellitus.
  Other Names: Amaryl
  Arms: Glimepiride

SUMMARY:
Patients with type 2 diabetes mellitus are exposed to an excessive heart failure risk secondary to left ventricular hypertrophy and impaired diastolic filling, a condition not addressed by currently available treatments. The abnormality results from obesity-induced volume overload, increased blood pressure, and myocardial fat accumulation. By improving metabolism, body weight, and blood pressure, Empagliflozin addresses the root causes of type 2 diabetes-associated myocardial disease. We will assess left ventricular mass, function, and lipid content in patients with type 2 diabetes mellitus using cardiac magnetic resonance imaging and spectroscopy as well as echocardiography before and after empagliflozin or glimepiride treatment. We expect to observe improvements in left ventricular mass, function, and fat content with empagliflozin. The results of the study will help to position empagliflozin as an antidiabetic agent with the added value of protecting the heart.

DETAILED DESCRIPTION:
Overview of Medical Indication Type 2 diabetes mellitus is associated with increased heart failure risk. The increased risk results in part from poor glycemic control and obesity, but concomitant arterial hypertension may also contribute. In the Framingham Heart Study, heart failure risk increased by 5% in men and by 7% in women with each 1 kg/m2 increment in body mass index (BMI). Compared with normal weight subjects, obese subjects had a doubling of heart failure risk. Given the rapid increase in the prevalence of obesity and type 2 diabetes mellitus, the number of heart failure patients is likely to increase sharply.

Evidence Heart failure in obesity is explained by increased left ventricular mass and impaired left ventricular diastolic filling rather than systolic dysfunction. Obesity is associated with volume expansion and increased cardiac output. Arterial blood pressure also increases with increasing obesity. In addition, type 2 diabetes mellitus may directly elicit abnormalities in myocardial metabolism and function through intramyocardial triglyceride deposition and lipotoxicity. In a study from our group, obese women with insulin resistance showed increased myocardial lipid accumulation compared with obese insulin-sensitive women, and intramyocardial lipids were reduced by dietary weight loss. Finally, intramyocardial lipids are associated with impaired diastolic function in patients with type 2 diabetes mellitus. Myocardial insulin resistance may also contribute to heart failure, because genetic deletion of cardiac insulin receptors in mice worsens catecholamine-mediated myocardial injury. Heart failure risk may be further exacerbated through obesity-induced neurohumoral activation and systemic inflammation. Inflammatory cytokines are elevated in heart failure and modulate cardiac remodelling through various mechanisms including myocardial hypertrophy, fibrosis, and apoptosis.

Sodium-glucose cotransporter 2 (SGLT2) inhibitors are a new drug class for the treatment of type 2 diabetes mellitus. SGLT2 inhibitors may be particularly suitable in improving cardiac structure and function because they substantially improve systemic glucose metabolism, lower blood pressure, and reduce body weight. These effects reduce sympathetic vasomotor tone, and renin-angiotensin-system activity. Thus, SGLT2 inhibitors including empagliflozin ameliorate metabolic and hemodynamic risk factors tightly linked with left ventricular hypertrophy and heart failure risk. Recently published outcome data suggest a beneficial effect of empagliflozin on heart failure hospitalisation rates and on overall cardiovascular mortality in patients with type 2 diabetes and previously diagnosed cardiovascular disease.

Study Rationale Patients with type 2 diabetes mellitus are exposed to an excessive heart failure risk secondary to left ventricular hypertrophy and impaired diastolic filling, a condition not addressed by currently available treatments. The abnormality results from obesity-induced volume overload, increased blood pressure, and myocardial fat accumulation. By improving metabolism, body weight, and blood pressure, empagliflozin addresses the root causes of myocardial disease associated with type 2 diabetes-. We will assess left ventricular mass, function, and lipid content in patients with type 2 diabetes mellitus before and after 24 weeks treatment with metformin plus empagliflozin or glimepiride. We expect to observe improvements in left ventricular mass, function, and fat content with empagliflozin. The results of the study will help to understand the mechanisms of cardioprotective effects of empagliflozin that have been revealed recently.

ELIGIBILITY:
Inclusion Criteria:

1. women and men ≥40 and <80 years of age
2. patients with type 2 diabetes mellitus on stable anti-diabetic treatment for the last 3 months; at screening the following treatment conditions are allowed:

   * metformin + sulfonylurea with HbA1c ≥6.5% and ≤9.0%
   * metformin monotherapy with HbA1c ≥7.5% and ≤ 9.0%
   * metformin + dipeptidylpeptidase-IV inhibitor with ≥6.5% and ≤9.0%
3. waist circumference ≥80 cm in women or ≥94 cm in men
4. office blood pressure ≤150/95 mm Hg with a stable dose of a maximum of 4 antihypertensive medications for the last 3 months (24h ambulatory blood pressure measurement (ABPM) is allowed to check accuracy of office values; inclusion with 24h mean blood pressure ≤145/90 mm Hg is possible)
5. women without childbearing potential defined by:

   * at least 6 weeks after surgical sterilization by bilateral tubal ligation or bilateral oophorectomy
   * hysterectomy
   * ≥ 50 years and in postmenopausal state > 1 year
   * < 50 years and in postmenopausal state > 1 year with serum follicle-stimulating Hormone (FSH) > 40 IU/l and serum estrogen < 30 ng/l or a negative estrogen test, both at screening
6. women of childbearing potential with a negative serum pregnancy test at screening who agree to meet one of the following criteria from the time of screening, during the study and for a period of 4 days following the last administration of study medication:

   * correct use of reliable contraception methods. The following are acceptable: hormonal contraceptives (combined oral contraceptives, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release), intrauterine device (IUD/IUS) or a double barrier method, e.g. condom and occlusive cap (diaphragm or cervical/vault caps) with spermicide (foam, gel, film, cream or suppository)
   * true abstinence (periodic abstinence and withdrawal are not acceptable methods of contraception)
   * sexual relationship only with female partners
   * sterile male partners
7. signed written informed consent and willingness to comply with treatment and follow-up
8. capability of understanding the investigational nature, potential risks and benefits of the clinical trial

Exclusion Criteria:

1. diabetes mellitus type 1
2. uncontrolled diabetes mellitus type 2 with fasting glucose > 13.3 mmol/l confirmed on a second day
3. previous treatment with insulin, glucagon-like peptide-1 analogues, or pioglitazone during the last year before screening
4. previous treatment with empagliflozin
5. acute illness at screening or randomization according to judgement by the investigator or patient
6. known or suspected hypersensitivity to empagliflozin, glimepiride or any excipients; known or suspected hypersensitivity to sulfonylureas or sulfonamides
7. history of multiple severe hypoglycemic episodes
8. any condition prohibiting MRI studies (e.g. metal implants, claustrophobia, body weight too high) including any suspected reaction after contrast agent application
9. patient actively attempted to lose weight or experienced unintentional clinically significant weight loss during the last 3 months
10. bariatric surgery or other gastrointestinal surgery procedures that induce chronic malabsorption
11. treatment with any weight loss drug in the preceding 6 months
12. planned significant changes of pre-study physical activity level during study participation
13. heart failure New York Heart Association (NYHA) III - IV
14. patients with known severe cardiovascular disease (e.g. myocardial infarction, unstable angina, stable coronary artery disease, stroke or transient ischemic attack)
15. calculated glomerular filtration rate (eGFR) <60 ml/min/1,73 m2
16. treatment with loop diuretics
17. chronic diarrhea, any clinical signs of volume depletion or a haematocrit > 48 % (women) and > 53 % (men)
18. history of severe volume depletion that required medical therapy
19. chronic lower urinary tract infections (but not simple asymptomatic bacteriuria)
20. known acute or chronic liver disease or screening liver enzymes > 3 x upper limit of normal (ULN)
21. serum potassium < 3.6 or > 5.0 mmol/l
22. glucose-6-phosphate dehydrogenase deficiency
23. anemia of unknown origin
24. pregnancy or lactation period
25. treatment with systemic glucocorticoids during the last 3 months before screening
26. chronic treatment with non-steroidal anti-inflammatory drugs (NSAIDs)
27. changes in thyroid hormone dosage (stable doses of thyroid hormones for the last 3 months are acceptable)
28. history of drug or alcohol abuse or current abuse
29. psychosomatic or psychiatric diseases requiring hospitalization during the last 12 months; ongoing treatment with one tricyclic or selective serotonin re-uptake Inhibitor (SSRI) antidepressant drug at a stable dose since the last 3 months is acceptable except for fluoxetine
30. medical history of cancer except for strictly localized tumors
31. any medical or surgical intervention planned for the next 7 months after randomization not allowing study participation according to the investigator´s judgment
32. current participation in any other clinical trial or participation in another clinical trial within 30 days before screening

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2017-09-27 (Actual)

PRIMARY OUTCOMES:
change in left ventricular mass | baseline and 24 weeks
  change in left ventricular mass determined by cardiac MRI as the difference between 24 weeks and baseline

SECONDARY OUTCOMES:
change in left ventricular end-systolic volume | baseline and 24 weeks
  change in left ventricular end-systolic volume (cMRI, 24 weeks - baseline)
change in left ventricular function | baseline and 24 weeks
  change in left ventricular function (cMRI, 24 weeks - baseline)
change in intramyocardial lipid content | baseline and 24 weeks
  change in intramyocardial lipid content (cMR spectroscopy, 24 weeks - baseline)
change in diastolic function | baseline and 24 weeks
  change in diastolic function (echocardiography, 24 weeks - baseline)
change in HbA1c | baseline and 24 weeks
  change in HbA1c (24 weeks - baseline)
change in fasting plasma glucose concentration | baseline and 24 weeks
  change in fasting plasma glucose concentration (24 weeks - baseline)
change in body weight | baseline and 24 weeks
  change in body weight (24 weeks - baseline)
change ambulatory blood pressure | baseline and 24 weeks
  change in ambulatory blood pressure (24 weeks - baseline)
change in left ventricular end-diastolic volume | baseline and 24 weeks
  change in left ventricular end-diastolic volume (cMRI, 24 weeks - baseline)
change in fasting serum insulin concentration | baseline and 24 weeks
  change in fasting serum insulin concentration (24 weeks - baseline)
change in waist circumference | baseline and 24 weeks
  change in waist circumference (24 weeks - baseline)
change in body fat mass | baseline and 24 weeks
  change in body fat mass (24 weeks - baseline)

OTHER OUTCOMES:
change in cardiac fibrosis | baseline and 24 weeks
  change in cardiac fibrosis (cMRI, 24 weeks - baseline)
change in global long strain | baseline and 24 weeks
  change in global long strain (echocardiography, 24 weeks - baseline)
number of participants with abnormal laboratory values in the blood | baseline and 4, 8, 12, 16, 20, 24 weeks
  To determine this number, blood electrolytes, blood count, hematocrit, liver function tests, blood urea and creatinine will be measured at baseline and every 4 weeks thereafter.
number of participants with abnormal laboratory values in the urine | baseline and 4, 8, 12, 16, 20, 24 weeks
  To determine this number, dip stick urine analysis will be performed at baseline and every 4 weeks thereafter (glucose will be measured but not reported to investigators to ensure blinding).
number of participants with lower urinary tract infections or genital fungal infections | baseline and 24 weeks
  To determine this number, signs and symptoms of lower urinary tract infections or genital fungal infections will be recorded at baseline and every 4 weeks thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Jordan, Prof. Dr., Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No